CLINICAL TRIAL: NCT00673712
Title: Phase 4 Multicenter Infection Surveillance Study Following Cardiac Surgical Procedures
Brief Title: Multicenter Infection Surveillance Study Following Open Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halyard Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iflocv2008
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2015-04

CONDITIONS: Surgery; Pneumonia; Surgical Site Infection
Keywords: Coronary Artery Bypass Graft Surgery; Pneumonia; Surgical Site Infection
MeSH Terms: conditions — Pneumonia; Surgical Wound Infection | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Sternal Block (Experimental): Continuous Sternal block with infusion of local anesthetic via ON-Q Painbuster Silver Soaker system
  Interventions: Device: Continuous Sternal Block
- Opioid based analgesia (Active Comparator): Opioid based analgesia including Patient controlled analgesia plus IM, Oral narcotics and other analgesics
  Interventions: Drug: Opioid based analgesia

INTERVENTIONS:
Device: Continuous Sternal Block — Elastomeric Pump for Continuous Infusion of Local Anesthetic
  Other Names: ON-Q; PainBuster
  Arms: Continuous Sternal Block
Drug: Opioid based analgesia — Opioid Analgesic agents delivered by:
  PCA on demand mode IV injections PRN IM injections PRN Oral PRN
  Other Names: PCA
  Arms: Opioid based analgesia

SUMMARY:
The main goals of the study are as follows: (1) to determine the correlation between pain management using continuous infusion of local anesthetics and the incidence of pneumonia and surgical infection in cardiac surgery patients; and (2) to evaluate the relationship between hospital-acquired pneumonia and surgical infection and patient outcomes, including length of hospital stay.

DETAILED DESCRIPTION:
Nosocomial infections are recognized as an important cause of increased patient morbidity and mortality. The reported prevalence for nosocomial infections most commonly ranges from 5 to 20%, but can be significantly greater among patients requiring intensive care. The most common sites of hospital acquired infection include the lung, urinary tract, surgical wounds, and the bloodstream. Patients undergoing cardiac surgery appear to be at increased risk for the development of nosocomial infections due to the presence of multiple surgical wounds (chest and lower extremity incisions), frequent postoperative utilization of invasive devices (i.e. central venous catheters, chest drains, intra-aortic balloon counter pulsation, pulmonary artery catheter), and the common use of prophylactic or empiric antibiotics in the perioperative period. In the cardiac surgical postoperative period, nosocomial infections have been found to be associated with prolonged length of stay (LOS) in the ICU and total hospitalization, development of multiorgan dysfunction, and increased hospital mortality. Nosocomial Pneumonia (NP) is in fact the leading cause of mortality due to hospital-acquired infections. Patients with Ventilator Associated Pneumonia (VAP) have been found in various studies to have significantly higher mortality rates than those without VAP, with ranges of 20.2-45.5% and 8.5-32.2%, respectively. Strategies that both reduce postoperative pain and sedation have the potential to reduce postoperative pneumonia by allowing earlier extubation and more effective pulmonary toilet post-extubation. Non-opioid pain management has the potential to reduce NP rates because of superior pain management, as well as the reduction in opioids required, and the concomitant avoidance of opioid side effects. The clinical and financial consequences of NP justify aggressively pursuing strategies aimed at prevention. Specifically, these strategies are targeted at reducing the incidence of NP by addressing the modifiable risk factors including prolonged endotracheal intubation and ventilator support, sedation, and long hospital LOS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, >18 years of age;
* Scheduled for elective cardiac surgical procedure, including coronary revasculari-zation or valve surgery;
* Provision of informed consent

Exclusion Criteria:

* Patients with a prior allergic reaction or dependency to morphine, Demerol, Di-laudid, Fentanyl, Marcaine (bupivacaine), lidocaine or Naropin (ropivacaine);
* Cardiac transplant patients
* Inability to perform follow-up assessments;
* Pre-existing infection (pneumonia or surgical site)
* Repeat of primary surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Husain, MD, Principal Investigator — The Cleveland Clinic
Locations (8):
- United States (8):
  - St. Vincents East, Birmingham, Alabama
  - Christianna Care Health System, Newark, Delaware
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Ochsner, New Orleans, Louisiana
  - Cape Fear valley Hospital, Fayetteville, North Carolina
  - Medcentral Hospital, Mansfield, Ohio
  - Methodist Hospital, Houston, Texas
  - Waukesha Medical Center, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Opioid Based Analgesia: Opioid based analgesia including Patient controlled analgesia plus IM, Oral narcotics and other analgesics
  Opioid based analgesia: Opioid Analgesic agents delivered by:
  PCA on demand mode IV injections PRN IM injections PRN Oral PRN
Period: Overall Study
Arm/Group | Continuous Sternal Block | Opioid Based Analgesia
Started | 321 | 326
Completed | 321 | 326
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Sternal Block | Opioid Based Analgesia | Total
Number analyzed (Participants) | 321 | 326 | 647
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12.1) | 65.2 (11.5) | 64.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 97 | 198
  Male | 220 | 229 | 449
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 26 | 55
  White | 273 | 277 | 550
  More than one race | 6 | 12 | 18
  Unknown or Not Reported | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 321 | 326 | 647

OUTCOME MEASURES:

1. Primary Outcome: Hospital Acquired Pneumonia
Description: Pneumonia diagnosed during hospitalization
Time Frame: 30 days postoperative
Population: all randomized subjects
Measure: Number; unit: participants
Arm/Group | Continuous Sternal Block | Opioid Based Analgesia
Number analyzed (Participants) | 321 | 326
participants | 8 | 18

2. Secondary Outcome: Surgical Site Infection
Description: surgical site infection diagnosed within 30 days post surgery
Time Frame: 30 days postoperative
Population: all randomized subjects
Measure: Number; unit: participants
Arm/Group | Continuous Sternal Block | Opioid Based Analgesia
Number analyzed (Participants) | 321 | 326
participants | 17 | 19

3. Secondary Outcome: Hospital Length of Stay
Description: time (days) from date of admission to discharge
Time Frame: primary admission
Population: all randomized subjects
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Continuous Sternal Block | Opioid Based Analgesia
Number analyzed (Participants) | 321 | 326
days | 8.8 (29.9) | 9.5 (29.6)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Continuous Sternal Block | Opioid Based Analgesia
Serious Adverse Events (participants affected / at risk) | 0/321 | 0/326
Other Adverse Events (participants affected / at risk) | 0/321 | 0/326

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No